CLINICAL TRIAL: NCT02654899
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess Safety, Tolerability, And Pharmacokinetics Of Single Escalating Oral Doses Of Pf-06815345, As Well As Characterize The Pharmacokinetics Of Two Formulations And Effect Of Food On Pharmacokinetics Of One Formulation Of Pf-06815345 Administered To Healthy Adult Subjects
Brief Title: Single Dose Study of PF-06815345 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial discontinued on 04Apr2016 as a strategic business decision not to pursue the indication. Decision to terminate not due to safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C0281001; 2015-003935-36 (EudraCT Number)
Record Dates: First submitted 2015-11-17; First posted 2016-01-13 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Hypercholesterolemia
Keywords: Healthy subjects; Single Ascending Dose; Hyperlipidemia; Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1_Cohort 1_Active; (Experimental): Single ascending dose of PF-06815345
  Interventions: Drug: PF-06815345
- Part 1_Cohort 1_Placebo; (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Part 1_Cohort 2_Active (Experimental): Single ascending dose of PF-06815345
  Interventions: Drug: PF-06815345
- Part 1_Cohort 2_Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Other: Placebo
- Part 2 (Experimental): Single dose of solid dosage formulation (test) versus liquid dosage formulation (reference) of PF-06815345
  Interventions: Drug: PF-06815345

INTERVENTIONS:
Drug: PF-06815345 — PF-06815345 will be administered as a liquid dosage formulation
  Arms: Part 1_Cohort 1_Active;; Part 1_Cohort 2_Active
Other: Placebo — Placebo
  Arms: Part 1_Cohort 1_Placebo;; Part 1_Cohort 2_Placebo
Drug: PF-06815345 — PF-06815345 will be administered as either solid dosage formulation or liquid dosage formulation
  Arms: Part 2

SUMMARY:
The current study is the first clinical trial proposed with PF-06815345. It is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) following administration of single oral doses of PF-06815345 to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and female of non-childbearing potential;
* Age of 18-55, inclusive;
* Body Mass Index 17.5-34.9 kg/m2, inclusive;
* Body weight >50 kg;
* Not on any prescription or non-prescription drugs within 7 days or 5 half-lives prior to first dose.

Exclusion Criteria:

- Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergises, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline (Day 0) up to 28 days after last dose of study medication
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06815345 | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] for PF-06815345 | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  AUC (0-infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Maximum Observed Plasma Concentration (Cmax) for PF-06815345 | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Concentration for PF-06815345 | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) for PF-06815345 | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Apparent Oral Clearance (CL/F) for PF-06815345 | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) for PF-06815345 | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for the metabolite (PF-06811701) | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] for metabolite (PF-06811701) | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  AUC (0-infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Maximum Observed Plasma Concentration (Cmax) for metabolite (PF-06811701) | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Concentration for metabolite (PF-06811701) | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Plasma Decay Half-Life (t1/2) for metabolite (PF-06811701) | 0, 0.5, 1, 2, 3, 4, 6, 10, 14, 24, and 48 hours post dose
  Plasma Decay Half-Life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0281001&StudyName=A%20Phase%201%2C%20Randomized%2C%20Double-blind%2C%20Placebo-controlled%20Study%20To%20Assess%20Safety%2C%20Tolerability%2C%20And%20Pharmacokinetics%20Of%20Single%20Escalating%20Oral%20Doses%20Of%20Pf-06815345%2C%20As%20Well%20As%20Characterize%20The%20Pharmacokinetics%20Of%20Two%20Formulations%20And%20Effect%20Of%20Food%20On%20Pharmacokinetics%20Of%20One%20Formulation%20Of%20Pf%E2%80%9106815345%20Administered%20To%20Healthy%20Adult%20Subjects